CLINICAL TRIAL: NCT00309543
Title: A Prospectively Randomized Study on Adjuvant Chemotherapy in Patients With Operated Colon Carcinoma Dukes B (Stage II; T3-4, N0, M0).
Brief Title: Randomized Trial on Adjuvant Chemotherapy in Colon Carcinoma Dukes B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG 91
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2006-03

CONDITIONS: Colon Cancer Stage II
Keywords: Fluorouracil; Leucovorin; Colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Fluorouracil
Drug: Leucovorin

SUMMARY:
This clinical investigation examined the influence of cytostatic chemotherapy with 5-fluorouracil, modulated by biologically active leucovorin, on patients' survival time following surgery for colon carcinoma Stage II.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically verified, operable colon carcinoma Stage II (RO, T3-4, N0, M0)
* Age: less than 80 years
* WHO Performance > 2
* Adequate bone marrow reserve, renal and hepatic functions
* Informed consent

Exclusion Criteria:

* Rectal cancer
* R1or R2 resection; carcinosis peritonei
* Start of treatment > 42 days postop; other adjuvant radiotherapy, chemotherapy or immunotherapy
* Serious concomitant disease, in particular chronically inflammatory large intestine, cardiopathic or metabolic disease, malignant second carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636
Dates: Start 1993-11

PRIMARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (18):
- Austria (18):
  - Hospital Guessing, Güssing, Burgenland
  - Hospital Oberpullendorf, Oberpullendorf, Burgenland
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - State Hospital Wolfsberg, Wolfsberg, Carinthia
  - Hospital Hainburg, Hainburg an der Donau, Lower Austria
  - Hospital Krems, Krems, Lower Austria
  - Hospital Tulln, Tulln, Lower Austria
  - Hospital Waidhofen/Thaya, Waidhofen A. D. Thaya, Lower Austria
  - Hospital Wiener Neustadt, Surgery, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University Salzburg - Oncology, Salzburg, Salzburg
  - Medical University of Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Leoben, Styria
  - Hospital St. Vinzenz, Zams, Tyrol
  - State Hospital Kirchdorf, Kirchdorf, Upper Austria
  - Hospital Kreuzschwestern Wels, Wels, Upper Austria
  - Medical University Vienna, General Hospital, Vienna, Vienna
  - Wilheminenspital, Internal Medicin I, Vienna, Vienna
  - State Hospital Feldkirch, Feldkirch, Vorarlberg

REFERENCES:
- See also: Related Info — http://www.abcsg.at